CLINICAL TRIAL: NCT02907788
Title: Inflammatory Markers in Broncho-alveolar Lavage Fluid as Risk Factors for Lung Disease in Infants With Cystic Fibrosis: the I-BALL Study
Acronym: I-BALL
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: Emory University (Other); UMC Utrecht (Other)
Responsible Party: Principal Investigator, Dr. H.M. Janssens, Dr, MD, PhD, Erasmus Medical Center
Other Study IDs: NL49725.078.14
Record Dates: First submitted 2016-09-06; First posted 2016-09-20 (Estimated); Last update posted 2021-11-05 (Actual); Status verified 2021-11

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; Neutrophils; PMN; Inflammation; Lung disease; PRAGMA
MeSH Terms: conditions — Cystic Fibrosis; Inflammation; Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — * Whole Blood
  * Bronchoscopies and bronchoalveolar lavage fluid (BALF)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cystic Fibrosis patients: Patient with cystic fibrosis diagnosed by Heel-prick screening
- non-CF patients: Children who undergo bronchoscopy for another reason, without CF: eg gastro-esophageal reflux.

SUMMARY:
Airway disease, featuring intense inflammation, is the main cause of morbidity and mortality in cystic fibrosis (CF). Mechanisms of CF airway inflammation remain unclear, hampering development of better treatments.This time-sensitive ancillary study leverages a unique longitudinal cohort of CF infants, assessing the early phase of airway disease. Through the use of innovative cell and fluid based tools for in vivo profiling and in vitro testing of BALF samples, this translational effort will yield unprecedented insights into mechanisms of PMN dysfunction in CF, and assess new paths for early intervention.

DETAILED DESCRIPTION:
Rationale: Airway disease, featuring early and intense inflammation and leading to progressive lung damage, is the main cause of morbidity and mortality in cystic fibrosis (CF). Mechanisms of CF airway inflammation remain unclear, hampering development of better treatments. Recent introduction of heel-prick screening for CF provides a unique longitudinal cohort of CF infants, in which the early phase of airway disease can be assessed. In our hospital the investigators set up a clinical protocol for monitoring these infants in a structured way, using chest computed tomography (CT) and bronchoscopies with collection of broncho-alveolar lavage fluid (BALF) to assess early lung damage. Our protocol is designed according to the protocol used by the Australian AREST-CF consortium. Preliminary data show that lipid profiles differ in BALF from CF infants with a high score for lung damage, compared with a low score (minimal lung damage). Some of these lipids are products of activated polymorphonuclear neutrophils (PMN's). Others are receptor-activating molecules involved in the resolution of inflammation and tissue injury. Also, in a pilot study, it was shown that CF airway PMNs are differently programmed than in normal airways, which leads to increased release of inflammatory factors and toxic enzymes. The hypothesize is that CFTR deficiency causes abnormal inflammatory signaling in the lung of CF infants, resulting in abnormal programming of infiltrating PMNs, and subsequently excessive and chronic lung disease.

Objectives: To better understand the progression of early CF lung disease the investigators aim to study lipid profiles and PMN dysfunction in relation to the severity of early lung disease in infants with CF, using BALF samples and peripheral blood. To optimally study these very precious samples, the investigators will make use of state-of-the-art technologies for in vivo profiling and in vitro testing of PMN function, including lipidomics and innovative cell- and fluid-based tools. Understanding the mechanisms at play in CF airway inflammation as it occurs in infants may lead to new paths for early intervention

Study design: Observational, exploratory in vitro study in BALF and peripheral blood from infants with CF, correlated with clinical data.

Study population: Children with CF diagnosed by heel-prick screening, who have a bronchoscopy and chest-CT for their annual check-up, at age 3 months (Utrecht),1, 3 or 5 years are eligible. Informed consent will be obtained from the parents.

Intervention: The bronchoscopy done to collect BALF is part of the routine clinical monitoring program. For this study, BALF that is not used for clinical testing will be used. Furthermore, venous puncture is performed for clinical routine blood tests, and one extra vial of EDTA blood will be drawn.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with CF, confirmed with 2 mutations found by genetic analysis, either from heel-prick screening or diagnosed later in life
* Aged 3 months (Utrecht),1, 3 or 5 years, who undergo bronchoscopy and chest CT scan as part of the routine monitoring program for CF
* Informed consent from parents

Exclusion Criteria:

* Absence of previously given informed consent for use of encoded clinical data for scientific purposes

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All CF patients enrolled in the AREST-CF program of the paediatric CF centre at Sophia Children's Hospital and Wilhelmina Children's Hospital.
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Lipid profiles with early lung disease in CF. | 5 years
  Lipidomics endpoints: The primary end-points are the different bioactive lipid levels in BALF of infants with CF using liquid chromatography (LC) coupled to Mass spectrometry (MS). Lipid profiles will be derived of the BALF supernatant
Surface markers of reprogrammed PMNs in BALF of infants with CF | 5 years
  Our primary endpoint for BALF cells flowcytometry analysis is surfacemarkers on airway PMNs (exocytosis of NE-rich granules), which was shown to correlate with lung function in chronic CF disease

SECONDARY OUTCOMES:
PRAGMA-CT scores of infants with CF | 5 years
  Secondary endpoints will include chest CT scores according to the PRAGMA scoring system

CONTACTS AND LOCATIONS:
Overall Officials: Rabindra Tirouvanziam, Assistant Professor, Principal Investigator — Emory University
Locations (1):
- Erasmus MC -Sophia childrens hospital, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No